CLINICAL TRIAL: NCT07015957
Title: Kupewa: Optimizing Implementation Strategies for Cervical Cancer Prevention
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other); Partners in Hope, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-FY2025-9686; 1U01CA294756 (NIH)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1: In-person training (Active Comparator)
  Interventions: Behavioral: In-person training
- Condition 2: In-person training + Prompt (Experimental)
  Interventions: Behavioral: In-person training; Behavioral: Prompts
- Condition 3: In-person training + Coaching (Experimental)
  Interventions: Behavioral: In-person training; Behavioral: Coaching
- Condition 4: In-person training + Prompt + Coaching (Experimental)
  Interventions: Behavioral: In-person training; Behavioral: Coaching; Behavioral: Prompts
- Condition 5: Virtual training (Experimental)
  Interventions: Behavioral: Virtual training
- Condition 6: Virtual training + Prompt (Experimental)
  Interventions: Behavioral: Virtual training; Behavioral: Prompts
- Condition 7: Virtual training + Coaching (Experimental)
  Interventions: Behavioral: Virtual training; Behavioral: Coaching
- Condition 8: Virtual training + Prompt + Coaching (Experimental)
  Interventions: Behavioral: Virtual training; Behavioral: Coaching; Behavioral: Prompts

INTERVENTIONS:
Behavioral: In-person training — An in-person educational session.
  Arms: Condition 1: In-person training; Condition 2: In-person training + Prompt; Condition 3: In-person training + Coaching; Condition 4: In-person training + Prompt + Coaching
Behavioral: Virtual training — A virtual educational session.
  Arms: Condition 5: Virtual training; Condition 6: Virtual training + Prompt; Condition 7: Virtual training + Coaching; Condition 8: Virtual training + Prompt + Coaching
Behavioral: Coaching — Short video vignettes plus reinforcing messages
  Arms: Condition 3: In-person training + Coaching; Condition 4: In-person training + Prompt + Coaching; Condition 7: Virtual training + Coaching; Condition 8: Virtual training + Prompt + Coaching
Behavioral: Prompts — Visual aide to remind providers to discuss cervical cancer prevention methods.
  Arms: Condition 2: In-person training + Prompt; Condition 4: In-person training + Prompt + Coaching; Condition 6: Virtual training + Prompt; Condition 8: Virtual training + Prompt + Coaching

SUMMARY:
The goal of this clinical trial is identify an effective and implementable set of implementation strategies to increase cervical cancer prevention in Malawi. The main questions it aims to answer are:

1. Which implementation strategies produce the greatest increase in provider recommendation for, and uptake of, cervical cancer prevention tools among people receiving HIV care.
2. What is the acceptability, appropriateness, feasibility, and cost of these implementation strategies.
3. What is the sustained effect of these implementation strategies. The implementation strategies will be conducted with health workers (clinical officers, nurses, and medical assistants): training, coaching, and a reminder system.

ELIGIBILITY:
Inclusion Criteria:

* Health workers: People who provide medical care and counseling (typically medical assistants, clinical officers, and nurses), and interact with adolescent girls and young women aged 9-24 and/or their parents/caregivers.
* Clients: Non-pregnant females aged 9-24 (for those aged 9-17, their male or female parent/guardian will also be eligible for participation) who present for HIV care at a participating health facility during the study period.

Exclusion Criteria:

* Health workers: Less than 18 years of age, or not an active and regular provider of medical care or counseling at the facility, or unable or unwilling to provide informed consent.
* Clients: <9 or >24 years old, or pregnancy, or unable or unwilling to provide informed consent.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Difference in prevalence of discussions surrounding methods of cervical cancer prevention | Months 7-18
  Discussions about methods of cervical cancer prevention will be reported by clients following each routine HIV care visit. This rate is defined as the percentage of visits during which there is a discussion about methods of cervical cancer prevention. This rate will be compared between the groups with and without each intervention component.

SECONDARY OUTCOMES:
Difference in prevalence of completing a cervical cancer prevention program | Months 7-18
  Completing a cervical cancer prevention program will be reported by clients following each routine HIV care visit. This prevalence is defined as the percentage of clients who complete a cervical cancer prevention program. This prevalence will be compared between the groups with and without each intervention component.
Difference in prevalence of initiating a cervical cancer prevention program among those uninitiated | Months 7-18
  This prevalence is defined among those who have not begun a cervical cancer prevention program at study entry. This prevalence will be compared between the groups with and without each intervention component.

OTHER OUTCOMES:
Acceptability of the implementation strategies | Months 1-9
  Health workers will be asked a set of questions to assess their perceived acceptability of the implementation strategies, based on the Theoretical Framework of Acceptability questionnaire, and these will be combined into an acceptability score (ranging from 0-27 with a higher score indicating greater acceptability). We will compare the average acceptability score between groups with and without each intervention component.

CONTACTS AND LOCATIONS:
Overall Officials: Corrina Moucheraud, Principal Investigator — New York University; Risa M Hoffman, Principal Investigator — University of California, Los Angeles; Sam Phiri, Principal Investigator — Partners in Hope, Inc.
Locations (1):
- Partners in Hope, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Fully deidentified survey data and focus group discussion transcripts
Supporting Information: Study Protocol, ICF
Access Criteria: Survey data will be deposited into a data repository after it has been fully de-identified. De-identified focus group discussion data will be available on a by-request basis via a data repository.

DOCUMENTS (6):
  • Informed Consent Form: Provider Baseline Consent English (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT07015957/ICF_000.pdf
  • Informed Consent Form: Parent Consent Baseline English (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT07015957/ICF_001.pdf
  • Informed Consent Form: Client Consent Baseline English (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT07015957/ICF_002.pdf
  • Informed Consent Form: Client Consent FollowUp English (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT07015957/ICF_003.pdf
  • Informed Consent Form: Parent Consent FollowUp English (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT07015957/ICF_004.pdf
  • Informed Consent Form: Provider FGD Consent English (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT07015957/ICF_005.pdf